CLINICAL TRIAL: NCT03154645
Title: Altitude Sickness Prevention With Ibuprofen Relative to Acetazolamide and Treatment Efficacy
Acronym: ASPIRATE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grant S Lipman (Other)
Responsible Party: Sponsor-Investigator, Grant S Lipman, Principal Investigator, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 40325
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Acute Mountain Sickness
MeSH Terms: conditions — Altitude Sickness | interventions — Ibuprofen; Acetazolamide

STUDY DESIGN:
Intervention Model Description: randomized double blind controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: visually identical pills
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ibuprofen (Active Comparator): ibuprofen, 600mg, three times a day, through to ascent to high altitude
  Interventions: Drug: Ibuprofen
- acetazolamide (Active Comparator): acetazolamide, 125mg, two times a day, through to ascent to high altitude
  Interventions: Drug: Acetazolamide

INTERVENTIONS:
Drug: Ibuprofen — non-steroidal anti-inflammatory drug
  Other Names: Motrin
  Arms: Ibuprofen
Drug: Acetazolamide — a diuretic
  Other Names: diamox
  Arms: acetazolamide

SUMMARY:
This double blind randomized trial will compare ibuprofen to acetazolamide for the prevention of acute mountain sickness. These drugs have never been directly compared for efficacy. The study population is hikers who are ascending at their own rate under their own power in a true hiking environment at the White Mountain Research Station, Owen Valley Lab (OVL) and Bancroft Station (BAR), Bancroft Peak, White Mountain, California.

DETAILED DESCRIPTION:
The specific aim of this study is to evaluate if acetazolamide will be similar to ibuprofen (i.e. Ibuprofen being non-inferior) in decreasing the incidence of Acute Mountain Sickness (AMS) in travelers to high altitude. It has been shown that ibuprofen taken 3 times a day 6 hours prior to ascent is effective for the prevention of AMS, with a number needed to treat of 4, decreasing the odds of getting AMS by a third. The efficacy appears to be similar to acetazolamide, with a NNT of 3 -8, although these two medications have not been directly compared in prevention of AMS. Acetazolamide is diuretic that is the only FDA approved AMS prophylactic medication and the most commonly used drug for AMS prevention. Although acetazolamide has been given a 1A indication, it has been shown to limit exercise capabilities at high altitude, and rapid ascent has been shown to attenuate its protective effects. Ibuprofen has been given a IIB recommendation by the Wilderness Medical Society Practice Guidelines, in part because it has not directly compared to acetazolamide. It is unknown if a non-steroidal anti-inflammatory can provide protection from AMS equivalent to acetazolamide.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 healthy non-pregnant volunteer
2. Sea-level dwelling (live at low elevation < 4000 ft)
3. Arrange your own transportation to WMRS (Bishop) by Friday evening of study weekend
4. Available for full study duration (Friday PM-Sunday AM)

Exclusion Criteria:

1. Age <18 or >65, Pregnant, Live at altitude >4000 ft
2. Slept at altitude > 4000ft within 1 week of study
3. Allergic to acetazolamide, sulfa drugs, or non-steroidal anti-inflammatories
4. Taking NSAIDs, Acetazolamide, or Corticosteroids 1 week prior to study
5. Medical History of Brain Tumor, increased brain pressure, pseudotumor cerebri, VP shunts, HACE, or HAPE.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-08-12 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
incidence of acute mountain sickness | 2 days
  incidence of acute mountain sickness by Lake Louise Questionnaire

SECONDARY OUTCOMES:
severity of acute mountain sickness | 2 days
  severity of acute mountain sickness by Lake Louise Questionnaire (0-15)
oxygen saturation | 2 days
  measurement of oxygen saturation (%) by fingertip pulse oximetry
Groningen Sleep Quality Questionnaire (GSQQ) | 2 days
  Groningen Sleep Quality Questionnaire (GSQQ) (0-14)

CONTACTS AND LOCATIONS:
Locations (1):
- White Mountain Research Station, Bishop, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Burns P, Lipman GS, Warner K, Jurkiewicz C, Phillips C, Sanders L, Soto M, Hackett P. Altitude Sickness Prevention with Ibuprofen Relative to Acetazolamide. Am J Med. 2019 Feb;132(2):247-251. doi: 10.1016/j.amjmed.2018.10.021. Epub 2018 Nov 10. PMID 30419226